CLINICAL TRIAL: NCT06908954
Title: A Phase I, Open-label, Parallel-group Study to Evaluate the Single-dose Pharmacokinetics of Palovarotene in Male and Female Participants With Moderate and Severe Hepatic Impairment and Matched Participants With Normal Hepatic Function
Brief Title: A Study of the Blood Levels of Palovarotene in Participants With Abnormal Liver Function Compared to Healthy Adult Participants After Intake of a Single Dose
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CLIN-60120-458
Record Dates: First submitted 2025-03-24; First posted 2025-04-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Hepatic Impairment; Healthy
MeSH Terms: interventions — Palovarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 Healthy participants (Experimental): Evaluation of the pharmacokinetics of IPN60120 in control healthy participants matching the age, sex and weight with hepatic impaired participants
  Interventions: Drug: Palovarotene
- Group 2 Moderate Hepatic impaired participants (Experimental): Evaluation of the pharmacokinetics of IPN60120 in Moderate Hepatic impaired participants (Child-Pugh class B)
  Interventions: Drug: Palovarotene
- Group 3 Severe Hepatic impaired participants (Experimental): Evaluation of the pharmacokinetics of IPN60120 in Severe Hepatic impaired participants (Child-Pugh class C)
  Interventions: Drug: Palovarotene

INTERVENTIONS:
Drug: Palovarotene — A single dose of maximum 10 mg of palovarotene will be administered orally on Day 1 to healthy control participants with normal hepatic function
  Arms: Group 1 Healthy participants
Drug: Palovarotene — A single 10 mg dose of palovarotene will be administered orally on Day 1 to Moderate hepatic impaired participants (Child-Pugh class B)
  Arms: Group 2 Moderate Hepatic impaired participants
Drug: Palovarotene — A single 10 mg dose of either 5 mg or 10 mg of palovarotene will be administered orally on Day 1 to Severe hepatic impaired participants (Child-Pugh class C).
  Arms: Group 3 Severe Hepatic impaired participants

SUMMARY:
The main aim of this study is to understand how moderate and severe liver impairment (based on the Child-Pugh classification) affects the body's processing of a single dose of 10 mg maximum of palovarotene, compared to healthy participants with normal liver function.

The study will also assess the safety and tolerability of the single dose of palovarotene.

Participants will be enrolled in stages and divided into three groups based on their liver function:

* Group 1: Healthy participants with normal liver function
* Group 2: Participants with moderate liver impairment
* Group 3: Participants with severe liver impairment (only enrolled if Group 2 results are safe and acceptable)

Blood samples will be taken to assess how the drug binds to proteins in the blood. Participants will undergo various safety checks and procedures. Participants will stay in the clinical unit until Day 5 for these assessments and will return on Day 10 for a final visit.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants must be 18 to 70 years of age (inclusive) at the time of signing informed consent.
* Body weight at least 60.0 kg with body mass index (BMI) within the range of 18.0 and 36.0 kg/m² (inclusive), at screening. BMI of >36.0 to ≤40.0 may be eligible if participant has moderate ascites scoring 3 points on the C-P criteria.
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical trials
* Clinical diagnosis of chronic hepatic disease (stable for more than 3 months) with a documented history of underlying hepatic insufficiency and no acute episodes of illness within 30 days prior to Day -1 (admission) and no significant change in disease status (i.e. up to 1 point in the C-P classification) from screening to Day -1.
* A stable medication regimen, defined as not starting new therapy(ies) or significant changing dosage(s) within 30 days prior to dosing.

Exclusion Criteria:

* Presence or significant history of cardiovascular, respiratory, hepatic (except for the hepatic impairment for those concerned), renal, gastrointestinal, biliary, mucocutaneous, endocrinological, haematological or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs, constituting a risk when taking the study intervention, or interfering with the interpretation of data.
* Lymphoma, leukaemia or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Breast cancer within the past 10 years.
* Use of any medications (prescription or over the counter), herbal tea, energy drinks (including natural stimulants), herbal products (e.g. St. John's wort, garlic, milk thistle) or supplements/supratherapeutic doses of vitamins within 14 days prior to Day 1 and through discharge, apart from those approved by the investigator and the sponsor's medical monitor. Those with hepatic impairment may take concomitant medications
* Use of any medications that are moderate or strong inhibitors or inducers of CYP3A4
* Donation or loss (excluding volume drawn at screening or during menses) of more than 250 mL of blood or blood product within 3 months prior to screening. In addition, plan of blood donation within 8 weeks after the last PK sampling.
* Presence of hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to the dose of study intervention.
* Positive hepatitis C antibody test result at screening or within 3 months prior to the dose of study intervention. Note: Participants with positive hepatitis C antibody due to prior resolved disease can be enrolled if a confirmatory negative hepatitis C ribonucleic acid (RNA) test is obtained.
* Positive hepatitis C RNA test result at screening or within 3 months prior to the dose of study intervention. Note: Test is optional and participants with negative hepatitis C antibody test are not required to also undergo hepatitis C RNA testing.
* Sensitivity to the study intervention, or components thereof (including inactive ingredients), or drug or other allergy that, in the opinion of the investigator (or medical monitor), contraindicates participation in the study
* Evidence of relevant active disease at screening, including gastroenterological (other than hepatic cirrhosis), cardiac (e.g. myocardial infarction in the past year, angina or congestive heart failure), renal, respiratory, haematological, neuropsychiatric or neoplastic (basal or squamous cell skin cancer is acceptable) disease.
* Acute hepatitis B (positive for HBsAg) or acute hepatitis C (positive for anti-hepatitis C virus (HCV) for a duration of less than 6 months). Note: Participants with chronic HCV (positive for HCV RNA or anti-HCV for more than 6 months) are eligible for enrolment, if stable, as assessed by the investigator.
* Primary sclerosing cholangitis or preliminary diagnosed biliary obstruction at screening.
* Current or chronic history of liver disease. This includes (but is not limited to hepatitis virus infections), drug- or alcohol-related liver disease, non-alcoholic steatohepatitis, autoimmune hepatitis, hemochromatosis, Wilson's disease, α-1 antitrypsin deficiency, primary biliary cholangitis, primary sclerosing cholangitis, or any other liver disease considered clinically significant by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2026-06-17 (Estimated); Study Completion 2026-06-17 (Estimated)

PRIMARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) | Over 96 hours postdose
  Measure of maximum observed plasma drug concentration (Cmax) (total and unbound) over 96 hours after dosing
Unbound fraction of drug in plasma (fu) | Over 96 hours postdose
  Measure of maximum observed plasma drug concentration (Cmax) (total and unbound) over 96 h after dosing
Time to maximum observed plasma concentration (Tmax) | Over 96 hours postdose
  Measure of AUC from time 0 to infinity (AUC0-∞) (total and unbound)
Area under the plasma concentration-time curve (AUC) from time 0 to infinity (AUC0-∞) | Over 96 hours postdose
  Measure of AUC from time 0 to infinity (AUC0-∞) (total and unbound)
AUC from 0 to time t corresponding to the last quantifiable concentration (AUC0-tlast) | Over 96 hours postdose
  Measure of AUC from 0 to time t corresponding to the last quantifiable concentration (AUC0-tlast) (total and unbound)
Apparent terminal elimination half life (T1/2) | Over 96 hours postdose
  Measure of apparent terminal elimination half-life over 96 hours post-dose
Apparent terminal elimination rate constant (λz). | Over 96 hours postdose
  Measure of apparent terminal elimination rate constant (λz) over 96 hours post-dose

SECONDARY OUTCOMES:
Percentage of participants with Adverse Events (AEs) | From Baseline to Day 10
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of Participants with clinically significant changes from baseline in Laboratory Parameters | At Day 2, Day 5 and Day 10
  Clinically significant change in laboratory parameters will be reported. The clinical significance will graded by the investigator.
Percentage of participants with clinically significant change from baseline in physical examinations | At Day 1, 2 and 3, Day 5 and Day 10
  Clinically significant changes in physical examinations will be reported. The clinical significance will be graded by the investigator.
Percentage of Participants With Clinically Significant Changes from baseline in Vital Signs | At Day 1, 2 and 3, Day 5 and Day 10
  Clinically significant changes in vital signs will be reported. The clinical significance will be graded by the investigator.
Percentage of participants with clinically significant change from baseline in 12-lead Electrocardiogram (ECG) readings | At Day 1, 2 and 3, Day 5 and Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (4):
- United States (4):
  - ERG - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - American Research Corporation/Texas Liver Institute, San Antonio, Texas
  - Pinnacle Clinical Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No